CLINICAL TRIAL: NCT05000125
Title: Comparison of the Hologic Genius Digital Diagnostics System With the ThinPrep Imaging System - a Retrospective Assessment
Brief Title: Comparison of the Hologic Genius Digital Diagnostics System With the ThinPrep Imaging System
Status: Completed | Type: Observational
Sponsor: Hologic Deutschland GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: BTS1702_21
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2021-08

CONDITIONS: Cervical Cancer Screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Slides from the German Co-Screening program: From 32506 LBC slides (ThinPrep, Hologic Inc., USA) from the German Co-screening program measured in 2020 with the TIS all abnormal findings according to Munich III groups (II-p - V) and 3% of normal slides (Munich III groups (I+II-a)) will be selected for the additional measurement with the Genius Digital cytology system.
  Interventions: Diagnostic Test: Hologic's Genius Digital Diagnostics System

INTERVENTIONS:
Diagnostic Test: Hologic's Genius Digital Diagnostics System — Genius Digital Diagnostics is a digital cytology platform to combine a new artificial intelligence (AI) algorithm with advanced volumetric imaging technology to help cytotechnologists and pathologists identify pre-cancerous lesions and cancer cells in women.

SUMMARY:
Quality assurance of the laboratory examinations. Retrospective non-interventional study with ThinPrep slides collected as part of the German Co-Screening Program for routine diagnostic. These slides will retrospectively be used to validate the Hologic Genius Digital Cytology (DC) system vs. the ThinPrep Imaging system (TIS).

DETAILED DESCRIPTION:
The cause of cervical cancer is a persistent infection with high-risk types of human papillomavirus (HPV). Cytology has been the gold standard for cervical screening since the introduction of routine screening with the Pap test in the 1950s due to its effect on mortality in regions with screening programs. Since that time, there have been several technological advances (LBC, Imaging) to improve and automate cervical cytology, resulting in increased disease detection and efficiency. The Hologic's Genius Digital Diagnostics System is a CE-IVD (CE-marked in vitro diagnostic device) marked digital cytology platform. For quality assurance and to retrospectively validate the Hologic Genius Digital Cytology (DC) system selected slides earlier measured with TIS will be additionally reviewed with the Genius Digital Diagnostic System in order to demonstrate clinical performance and efficiency.

Hologic's Digital Image Analysis Algorithm uses AI to identify diagnostically relevant objects of interest.Only anonymized results will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* LBC ThinPrep® samples are collected by gynaecologists and sent routinely to cytology laboratory CytoMol as part of the German Cervical cancer screening program.

Ages: 35 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Humans with a cervix.
Study Population: As part of the German National Cancer Plan, women over the age of 35 years will be given a cotest comprising a Pap smear and an HPV test, every three years.
Sampling Method: Probability Sample
Enrollment: 1994 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of detection of pre-cancerous lesions using Hologic Genius Digital Cytology Imaging scanner | 3 months
  To demonstrate non-inferiority, the appropriate approximative one sided 95% confidence interval for the true difference between the two approaches (Digital Cytology and the ThinPrep Imaging system (TIS)) will be constructed.

SECONDARY OUTCOMES:
Change in time needed to screen 80 slides using Hologic Genius Digital Cytology Imaging scanner. | 3 months
  To assess the impact on the workflow of the introduction of a Digital Cytology procedure to a high-throughput screening lab in Germany.
Clinical performance of Hologic Genius Digital Cytology Imaging scanner using cells on a ThinPrep® slide. | 3 months
  The performance of Hologic Genius Digital Cytology Imaging scanner during cervical cancer screening (using histology as reference method) will be assessed via sensitivity, specificity, positive and negative predictive values.

CONTACTS AND LOCATIONS:
Locations (1):
- CytoMol - MVZ für Zytologie und Molekularbiologie Frankfurt GbR, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No